CLINICAL TRIAL: NCT04605120
Title: Prospective, Non-randomized, Single Center Clinical Study of Cervical Interbody Fusion Using a Viral-inactivated Allogeneic Graft
Brief Title: Allogeinic Bone Paste
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biobank (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID-RCB : 2019-A02979-48
Record Dates: First submitted 2020-10-22; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Cervical Fusion; Cervical Disc Degeneration; Spinal Fusion
MeSH Terms: conditions — Klippel-Feil Syndrome

STUDY DESIGN:
Intervention Model Description: Non-randomized, Single centre
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeinic Bone Paste (Experimental): Supercritical CO2 viral-inactivated allogeinic bone paste derived from human living donor femoral heads
  Interventions: Procedure: Cervical fusion

INTERVENTIONS:
Procedure: Cervical fusion — 1- or 2-level ACDF (Anterior Cervical Discectomy and Fusion) combined with bone graft

SUMMARY:
This is a prospective, single arm, single center clinical study to evaluate efficacy and safety of a Supercritical CO2 viral-inactivated allogenic bone paste in cervical interbody fusion. Patient eligible for 1- or 2-level ACDF (Anterior Cervical Discectomy and Fusion) combined with bone graft after failure of well-conducted medical treatment will be screened for the study.

DETAILED DESCRIPTION:
Cervical and lumbar fusion are often the best option for various degenerative conditions that do not respond to conservative treatment. Historically, the reference technique for cervical fusion was the use of iliac crest autogenic bone graft (ICBG). However, the use of ICBG has several drawbacks, including the morbidity of the donor site, the increase in operating time and the variable quality of autograft. Alternatives to ICBG for cervical fusion include the use of allografts, graft extensions and osteobiological materials to improve fusion rates.

This is a prospective, single arm, single center clinical study to evaluate efficacy and safety of a Supercritical CO2 viral-inactivated allogenic bone paste in cervical interbody fusion. Patient eligible for 1- or 2-level ACDF (Anterior Cervical Discectomy and Fusion) combined with bone graft after failure of well-conducted medical treatment will be screened for the study.

Subjects will be followed up postoperatively per standard of care at 3 months, 6 months, 12 and 24 months at the clinic. The following outcomes will be measured: overall success, Neck Disability Index (NDI), VAS neck and arm pain, SF-12 health survey, major complications, subsequent surgery rate, and fusion rate on radiological examinations. The primary endpoint is a FDA composite definition of success comprising clinical improvement and absence of major complications and secondary surgery events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years old
2. Patient eligible for anterior cervical fusion combined with bone graft after failure of well-conducted medical treatment.
3. Arthrodesis performed on up to 2 levels and fused by one or more plates with an interbody cage on at least one level
4. Radicular signs and symptoms in one or both arms (i.e., pain, paresthesia, or paresis in a specific nerve root distribution) or symptoms and signs of acute or chronic myelopathy
5. X-ray diagnosis of cervical herniated disc and/or osteophyte at 1 or 2 levels depending on clinical signs and symptoms, disc degeneration, trauma without neurological damage
6. Ability and willingness to comply with project requirements
7. Written informed consent given by the subject or the subject's legally authorized representative

Exclusion Criteria:

1. Acute local or systemic infection
2. Women who are pregnant or in a desire to be pregnant or breast-feeding
3. Any contraindication to the proposed surgical procedure
4. Previous cervical surgery (either anterior or posterior)
5. Surgery performed over several operating times
6. Arthrodesis performed posteriorly or involving more than 2 levels or not requiring the use of a bone graft
7. Systemic disease, metabolic bone disease and autoimmune disease.
8. Use of any known drug to potentially interfere with the healing of bones and soft tissues (corticosteroids or immunosuppressive agents...)
9. Any other concomitant medical disease or treatment that could significantly alter the normal healing process as assessed by the investigator
10. Neoplasm of the spine
11. Severe mental or psychiatric disorders
12. Any other condition that, in the investigator's view, would adversely affect patient safety or would not meet the requirements of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall subject study success | 3, 6,12 and 24 months
  * Change from baseline Neck Disability Index (NDI): Patients will be evaluated preoperatively, at 3 months, 6 months, 12 and 24 months
  * Rate of Adverse Events (AEs) and Serious Adverse Events (SAEs) and reoperations during Follow-up visits
  * Interbody fusion rate measured by CT scans and standard radiographs at 3 months, 6 months, 12 and 24 months
  Overall subject study success is defined as (1) no device or implantation procedure related SAEs; (2) no additional surgical intervention at the operative level, including supplemental fixation, revision, and/or device removal; and (3) minimum 15-point improvement in NDI scores.

SECONDARY OUTCOMES:
Pain and Self reported outcomes | 3, 6, 12 and 24 months
  * Change from baseline neck and arm pain measured by Visual Analogue Scale (VAS): Patients will be evaluated preoperatively, at 3 months, 6 months, 12 and 24 months
  * Change from baseline Health Survey measured by SF-12: Patients will be evaluated preoperatively, at 3 months, 6 months, 12 and 24 months
  * Potential product benefits assessment by:
    * Surgery time (from incision to wound closure)
    * Product ease of use measured by Visual Analogue Scale (VAS) at immediate postoperative visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles LE HUEC, M.D., Prof, Principal Investigator — Polyclinique Bordeaux Nord Aquitaine - BORDEAUX - FRANCE
Locations (1):
- Polyclinique Bordeaux Nord Aquitaine, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No